CLINICAL TRIAL: NCT03410563
Title: The Analgesic Effect of Auditory Inputs and Its Relation to Psychological and Neurobiological Mechanisms
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: UAarhus_Sigrid
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-01

CONDITIONS: Analgesia
Keywords: Pain; Auditory inputs
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants
  Interventions: Behavioral: Auditory inputs

INTERVENTIONS:
Behavioral: Auditory inputs — Three different auditory inputs

SUMMARY:
The study investigates the analgesic effect of different auditory inputs. Employing a within-subject design, the study includes healthy participants that are exposed to thermal stimuli while listening to three different auditory inputs. By repeating this on separate test days, the involvement of bodily processes is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with normal hearing

Exclusion Criteria:

* Chronic pain conditions
* Other medical, psychiatric or neurological disorders
* Use of pain-relieving medication 24 hours prior to testing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scales | An average of 3 weeks (Participants are tested at three different test days across an average of 3 weeks; the primary outcome measure will be assessed after each thermal stimulus at the three test days)
  Acute pain assessed on visual analogue scales (0-100) examining pain intensity and pain unpleasantness

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology and Behavioural Sciences, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lunde SJ, Vuust P, Garza-Villarreal EA, Kirsch I, Moller A, Vase L. Music-Induced Analgesia in Healthy Participants Is Associated With Expected Pain Levels but Not Opioid or Dopamine-Dependent Mechanisms. Front Pain Res (Lausanne). 2022 Apr 4;3:734999. doi: 10.3389/fpain.2022.734999. eCollection 2022. PMID 35445208